CLINICAL TRIAL: NCT00274235
Title: Intermittent Preventive Treatment During Pregnancy in Benin: a Randomized, Open, and Equivalent Trial Comparing Sulfadoxine-Pyrimethamine With Mefloquine
Brief Title: Intermittent Preventive Treatment During Pregnancy in Benin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Institut de Recherche pour le Developpement (Other Government)
Collaborators: National Malaria Control Program, Benin (Other Government); Ministry of Foreign Affairs, France (Other Government); Institut des Sciences Biomédicales Appliquées, Bénin (Unknown); Faculté des Sciences de la Santé, Bénin (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UR10_01_2005
Record Dates: First submitted 2006-01-09; First posted 2006-01-10 (Estimated); Last update posted 2008-10-31 (Estimated); Status verified 2008-10

CONDITIONS: Malaria
Keywords: Malaria; Prevention; Pregnancy; Low birthweight; Anemia; Africa
MeSH Terms: conditions — Malaria; Anemia | interventions — mefloquine-sulfadoxine-pyrimethamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: sulfadoxine-pyrimethamine / mefloquine

SUMMARY:
Malaria in pregnancy is one of the most important preventable causes of low birthweight worlwide and a major cause of severe maternal anaemia contributing to maternal mortality. Intermittent Preventive Treatment (IPT) with sulfadoxine-pyrimethamine (SP) is the currently adopted government recommendation for malaria control during pregnancy in Benin, but the emergence and the spread of resistance to SP justifies the evaluation of alternative anti-malarial drugs. Mefloquine (MQ), which has been proven effective and reasonably safe in this indication, may be an interesting alternative to SP. The aim of this trial is to compare the efficacy and safety of sulfadoxine-pyrimethamine and mefloquine for IPT. It is an equivalent study designed to test the hypothesis that MQ is as efficacious as SP to prevent malaria in pregnancy, and that it could replace SP when resistance of Plasmodium falciparum becomes too elevated. Primary endpoint will be the proportion of infants with low birthweight. Secondary endpoints will be the proportion of mothers with placental plasmodial infection, and the proportion of mothers with anaemia at delivery.

DETAILED DESCRIPTION:
The trial will be conducted in two maternity clinics in Ouidah, 40km from Cotonou. A total of 1600 women will be selected and randomised to receive either SP (1500 mg sulfadoxine with 75 mg pyrimethamine) or MQ (15 mg/kg) twice during pregnancy at ante-natal clinic (ANC) visits. The first dose will be given between 16 and 28 weeks of gestation, the second between 30 and 36 weeks, and at least one month after the first dose. Women will be visited at home within one week after the initial and subsequent ANC visits to check for adverse reactions due to the study drugs. Peripheral blood samples will be collected on each ANC visit to assess for haemoglobin level and parasitemia. Peripheral, placental, and cord blood samples will be collected at delivery for haematological determinations and parasitological examination. Birthweight will be recorded and the gestational age assessed by the Ballard method. The mother and her child will be assessed for general health status six weeks after birth.

ELIGIBILITY:
Inclusion Criteria:

* Pregnancy between 16 and 28 weeks of gestation
* Residence near the maternity clinics
* Intention to continue the ante-natal care and deliver at the study maternity clinic
* Ability to take drugs by oral route
* Written informed consent (parents or guardian if aged < 18 years)

Exclusion Criteria:

* Pregnancy prior to 16 weeks or after 28 weeks of gestation
* Previous suspected reaction to sulfadoxine-pyrimethamine or mefloquine
* History of neurological or psychiatric event
* Intake of sulfadoxine-pyrimethamine or mefloquine within 4 weeks of enrollment
* Current treatment with halofantrine

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1600 (Estimated)
Dates: Start 2005-07; Primary Completion 2008-03 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
proportion of infants with low birthweight (<2,500 grams)

SECONDARY OUTCOMES:
mean birthweight
proportion of mothers with placental plasmodial infection
proportion of preterm deliveries
proportion of mothers with anaemia (Haemoglobin level (Hb)<11g/dl) and severe anaemia (Hb<8g/dl) at delivery
proportion of mothers with parasitaemia at delivery
proportion of adverse events after taking study drugs
proportion of congenital abnormalities
proportion of stillbirths

CONTACTS AND LOCATIONS:
Overall Officials: Michel Cot, MD, Principal Investigator — Institut de Recherche pour le Developpement
Locations (1):
- Institut de Recherche pour le Développement, Cotonou, Benin

REFERENCES:
- [Derived] Briand V, Bottero J, Noel H, Masse V, Cordel H, Guerra J, Kossou H, Fayomi B, Ayemonna P, Fievet N, Massougbodji A, Cot M. Intermittent treatment for the prevention of malaria during pregnancy in Benin: a randomized, open-label equivalence trial comparing sulfadoxine-pyrimethamine with mefloquine. J Infect Dis. 2009 Sep 15;200(6):991-1001. doi: 10.1086/605474. PMID 19656069
- [Derived] Briand V, Denoeud L, Massougbodji A, Cot M. Efficacy of intermittent preventive treatment versus chloroquine prophylaxis to prevent malaria during pregnancy in Benin. J Infect Dis. 2008 Aug 15;198(4):594-601. doi: 10.1086/590114. PMID 18598190